CLINICAL TRIAL: NCT03342820
Title: Impact of Muscular Fatigability on Spastic Co-contractions Between the Quadriceps and Hamstrings in Stroke Patients
Brief Title: Impact of Muscular Fatigability on Spastic Co-contractions After Stroke Patients
Acronym: COCON
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2016_50; 2017_A01605-48 (Other: ID-RCB number, ANSM)
Record Dates: First submitted 2017-10-16; First posted 2017-11-17 (Actual); Last update posted 2020-03-26 (Actual); Status verified 2020-03

CONDITIONS: Stroke; Spasticity, Muscle; Muscle Fatigue; Gait, Hemiplegic
MeSH Terms: conditions — Stroke; Muscle Spasticity; Gait Disorders, Neurologic | interventions — Muscle Fatigue

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Quadriceps muscle fatigue (Experimental): Quadriceps muscle fatigue
  Interventions: Procedure: Muscle fatigue

INTERVENTIONS:
Procedure: Muscle fatigue — Isokinetic quadriceps muscle fatigue of the paretic lower limb

SUMMARY:
This study evaluates the effects of an isokinetic fatigue protocol of the quadriceps on the amount of co-contractions of this last with the hamstrings during a maximal isometric flexion movement in hemiparetic stroke patients.

The effect of such a protocol on gait parameters and spasticity of the quadriceps will be evaluated also.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 80y
* Hemiparesis after a first-ever stroke > 3 months
* Spasticity of the quadriceps muscle
* Quadriceps strength at least at 3/5 (MRC testing)
* Subject able to walk at least 2min without rest
* Informed consent
* Social security affiliation

Exclusion Criteria:

* Severe comprehension troubles (language, cognitive or psychiatric disorders)
* History of previous stroke, locomotor or other neurological disorders
* Locomotor troubles affecting the paretic arm
* Contraindication to efforts : cardiac insufficiency, severe aortic valvular stenosis, recent heart failure, non treated high blood pressure, severe peripheral arterial disease
* Pregnancy or breastfeeding
* Adult subject to guardianship

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2018-01-19 (Actual); Primary Completion 2019-10-10 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Cocontraction Index (CCI) between the rectus femoris and the semitendinosus | one day
  ratio of the RMS of a the rectus femoris when acting as antagonist to the effort intended (knee flexion) to the RMS of the same muscle when acting as an agonist during a reciprocal maximal isometric knee flexion effort (500 ms around the peak of rectified EMG

SECONDARY OUTCOMES:
Cocontraction Index (CCI) between the other parts of the quadriceps and the semitendinosus muscle | one day
  ratio of the RMS of a the vastus medialis, lateralis and intermedius when acting as antagonist to the effort intended (knee flexion) to the RMS of the same muscle when acting as an agonist during a reciprocal maximal isometric knee flexion effort (500 ms around the peak of rectified EMG
Agonist Recruitment Index of the semitendinosus | one day
  ratio of the RMS of a muscle acting as an agonist during a given period to its largest RMS value observed during the 500 ms around its agonist recruitment peak
Isometric peak knee flexion torque | one day
  Isometric peak knee flexion torque assessed by a CONTREX dynamometer
Spasticity of the quadriceps | one day
  Tardieu scale angle
spatio-temporal gait parameters at comfortable speed | one day
  Gait speed
spatio-temporal gait parameters at comfortable speed | one day
  Gait cadence
spatio-temporal gait parameters at comfortable speed | one day
  Step length
Isometric peak knee extension torque | one day
  Isometric peak knee extension torque assessed by a CONTREX dynamometer
10 metre walk test (10MWT) | one day
  Assessment of max gait speed
2 minute walk test (2MWT) | one day
  Assessment of max walking endurance
perceived exertion at the end of the 2MWT (Borg Scale 6-20) | one day

CONTACTS AND LOCATIONS:
Overall Officials: Etienne Allart, Md, Principal Investigator — University Hospital, Lille
Locations (1):
- Hôpital Swynghedauw, CHU, Lille, France